CLINICAL TRIAL: NCT03768557
Title: The Effect of Acute Minocycline Administration on Emotional Processing and Cognition in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R50651/RE001
Record Dates: First submitted 2018-11-22; First posted 2018-12-07 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-11

CONDITIONS: Mood; Cognitive Change
MeSH Terms: interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minocycline (Experimental): single dose of minocycline (200mg)
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): lactose pills (400mg)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Minocycline — Minocycline (200mg)
  Arms: Minocycline
Other: placebo — Lactose (400mg)
  Arms: Placebo

SUMMARY:
There is growing interest in the possibility of producing more effective antidepressant treatments that target a wider range of pathways involved in depression, including anti-inflammatory and anti-glutamatergic systems. Minocycline is a novel pharmacological agent; in addition to its antibiotic and anti-inflammatory properties, it also acts in the brain as an anti-glutamatergic and anti-oxidant agent. Since both excessive glutamate and oxidative stress are implicated in major depression, and appear to be connected to pro-inflammatory activity, this drug offers a unique tool with which the investigators can measure the effects of targeting these pathways on emotional processing. Participants will receive a single dose of either the drug (200 mg minocycline) or placebo, and will then undergo a well-validated computerised battery of emotional processing tasks that have previously been shown to be sensitive to standard antidepressant drugs. Tasks include presentation of positive and negative emotional words or pictures, to which participants' responses are measured. These tasks have been widely used previously without any adverse effects.

DETAILED DESCRIPTION:
Current antidepressant treatments, which largely target monoamine pathways, are efficacious in treating many aspects of major depression, however it is estimated that more than 30% of depressed patients fail to respond to standard antidepressant medications. Thus, there is a strong clinical need to identify and investigate novel treatment strategies that target different pathways involved in the pathophysiology of mood disorders. Mounting evidence indicates a potentially important role of inflammation in major depression; both clinical and animal studies have shown that pro-inflammatory cytokines can induce a behavioural repertoire of symptoms collectively referred to as 'sickness behaviours,' which include cognitive and mood symptoms, such as depression, anxiety, memory impairment, fatigue and anhedonia. Furthermore, elevated levels of peripheral pro-inflammatory cytokines, such as tumour necrosis factor (TNF)-α and interleukin (IL)-6, have been consistently reported in clinical mood disorders, including major depression. Evidence also points to the ability of pro-inflammatory cytokines to cause excitotoxicity (due to increased release of glutamate) and oxidative stress that are strongly implicated in the pathophysiology of major depression. Such evidence has therefore led to growing interest in testing effects of anti-inflammatory treatments on mood and emotional function to investigate whether the inflammatory-mood pathway could represent a novel drug target for new antidepressant therapies.

Minocycline has been selected for use in the present study as it is a pharmacologically interesting agent with an unusual combination of anti-inflammatory activity, in addition to anti-glutamatergic, anti-oxidant and neuro-protective actions. Thus, owing to its central action on systems that are thought to be involved in major depression, minocycline provides an interesting tool to investigate effects on cognition and emotional processing, particularly negative affective biases.

Negative affective biases in emotional processing are highly relevant to clinical mood disorders and they are well-recognised in the aetiology and maintenance of depression, such that depressed individuals are more likely to interpret, focus on and remember negative compared to positive emotional cues in self-relevant neuropsychological tasks. Antidepressant treatments have been shown to cause early, subconscious positive changes in emotional processing biases, which are evident in computerised tasks after one single dose of antidepressant. Recent theory suggests that over time this positive change in emotional bias contributes to improved mood.

Since elevated inflammatory markers appear to negatively affect mood and neuropsychological function, the investigators believe there is a need to expand our understanding of the psychological effects of reducing inflammatory markers. To do so, subjects will be administered either a single dose of 200 mg minocycline or placebo, after which they will complete a well-validated computerized battery of psychological tasks, which includes paradigms such as facial expression recognition, emotional categorization and emotional memory tasks that have previously been shown to be sensitive to conventional antidepressant treatments in healthy volunteers.

The results of this study will be compared to effects of common antidepressant treatments found using this same model within the investigators' lab and others. If effects are found to be comparable, this could not only provide further support for the emotional processing theory of antidepressant action, but it could also help to identify novel therapeutic targets for new treatments that could benefit depressed patients who do not respond successfully to current antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* Participants are willing and able to give informed consent for participation in the study
* Male or female, aged between 18 and 55
* Body mass index (BMI) within the range of 19 - 30 kg/m2
* Sufficiently fluent in English to understand the tasks and instructions
* Female subjects must be outside of their pre-menstrual week on the testing day

Exclusion Criteria:

* Current or past history of any psychiatric disorder (e.g. depression, anxiety)
* Any medical contra-indication (for example hepatic impairment)
* Current use of any medication which, in the opinion of the study physician, will interfere with minocycline or cause any contraindications
* Known hypersensitivity to tetracyclines or to any of the excipients in minocycline capsules
* Steroidal or non-steroidal anti-inflammatory medication within preceding 2 weeks, including aspirin and ibuprofen
* Congenital or acquired immune deficiency (including participants receiving immunosuppressive or antimitotic drugs)
* Current pregnancy or breastfeeding
* Current substance misuse
* Recent (< 3 months) use of psychotropic drugs
* Participant in a psychological or medical study involving the use of medication within the last 3 months
* Participant in another study using the same / a similar battery of cognitive / emotional tasks in the last 3 months
* Current smoker of more than 5 cigarettes per day
* Dyslexia (given the nature of the computer tasks)
* Lactose intolerance (placebo is composed of lactose capsules)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Facial Expression Recognition Task | 2 hours
Emotional Categorization Task | 2 hours
Emotional Recall Task | 2 hours
Emotional Recognition Memory Task | 2 hours
Attentional Dot-Probe | 2 hours

SECONDARY OUTCOMES:
N-back Task | 2 hours
Contextual Cueing Task | 2 hours
Priming Task | 2 hours

OTHER OUTCOMES:
Concentration of the inflammatory marker TNF-alpha in serum Serum inflammatory cytokines and metabolites | 0 and 4 hours
Concentration of the inflammatory marker IL-6 in serum | 0 and 4 hours
Concentration of the inflammatory marker C-reactive protein in serum | 0 and 4 hours
Concentration of the stress hormone cortisol in serum | 0 and 4hours
Concentration of metabolites (amino acids and lipids) in serum | 0 and 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Warneford Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No